CLINICAL TRIAL: NCT02696369
Title: A Multi-center, Randomized, Double-blind, Crossover, phase4 Trial to Evaluate the Efficacy on Local Anesthesia and Safety of 2% Lidocaine HCl With Different Epinephrine Concentration in Patients Undergoing Surgical Extraction of Impacted Lower Third Molars
Brief Title: Trial to Evaluate the Efficacy on Local Anesthesia and Safety of 2% Lidocaine HCl With Different Epinephrine Concentration in Patients Undergoing Surgical Extraction of Impacted Lower Third Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HU-015
Record Dates: First submitted 2016-02-24; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Third Molar
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 2% Lidocaine HCL:Epinephrine inj. (Experimental): 2% Lidocaine HCL with epinephrine 1:200,000
  Interventions: Drug: 2% lidocaine HCl with epinephrine 1:200,000
- 2% Lidocaine HCL:Epinephrine inj. (3M) (Active Comparator): 2% Lidocaine HCl with epinephrine 1:80,000
  Interventions: Drug: 2% lidocaine HCl with epinephrine 1:80,000

INTERVENTIONS:
Drug: 2% lidocaine HCl with epinephrine 1:200,000
  Arms: 2% Lidocaine HCL:Epinephrine inj.
Drug: 2% lidocaine HCl with epinephrine 1:80,000
  Arms: 2% Lidocaine HCL:Epinephrine inj. (3M)

SUMMARY:
This study is Phase 4 trial which evaluates the safety and efficacy of 2% Lidocaine HCl with different epinephrine concentration in patients undergoing surgical extraction of impacted lower third molars

ELIGIBILITY:
Inclusion Criteria:

* Age over 19
* Physical grade 1 or 2 by American Society of Anesthesiologists (ASA)
* Mesioangular or horizontal angulation categorized by winter classification

Exclusion Criteria:

* Allergy or hypersensitivity about the investigated products
* Any infection or edema during the extraction
* The following patients: clotting disorder, hyperthyroidism, arteriosclerosis, cardiac insufficiency, other cardiovascular disorders
* Pregnancy or breast-feeding
* Any conditions that the investigator considers not to appropriate for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain visual analogue scale (VAS) | Immediately after the extraction
  To acess the pain immediately after the surgical extraction of impacted lower third molars

SECONDARY OUTCOMES:
Onset time of anesthesia | Immediately after administration of IP
Local anesthetic duration | Immediately after onset of anesthesia
Pain VAS | 2, 4, 6 hours after administration of the investigational product (IP)
Onset time of pain after administration of IP | Immediately after injection
Bleeding after extraction measured by the operator | Immediately after extraction
Questionnaire of satisfaction level of the operator | Immediately after extraction
Questionnaire of satisfaction level of the subjects | Immediately after extraction
Dosage of administrated IP | immediately after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Ansan, Kyeonggi-do, South Korea